CLINICAL TRIAL: NCT03932188
Title: Brain Imaging in Early Psychosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201904060
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse)
Keywords: early psychosis; prodrome; schizophrenia; psychosis
MeSH Terms: conditions — Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders; Schizophrenia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Individuals between 13-25 years old that do not meet criteria for any prodromal syndrome, any current or past psychotic disorder, or Cluster A personality disorder diagnosis
  Interventions: Behavioral: Mental Health Assessments and Computerized Cognitive Test; Device: MRI scan
- Prodromal/Early psychosis: Individuals between 13-25 years old that meet diagnostic criteria for a prodromal syndrome or early psychosis
  Interventions: Behavioral: Mental Health Assessments and Computerized Cognitive Test; Device: MRI scan

INTERVENTIONS:
Behavioral: Mental Health Assessments and Computerized Cognitive Test — Participants will be asked to complete questionnaires and will be asked questions that address a broad range of personal life experiences involving social, occupational, domestic, and other behaviors.
Device: MRI scan — Up to two MRI scan sessions will be done, altogether totaling just under 3 hours of scanning. MR scanners measure brain anatomy and activity using very strong magnets. No X-rays or radiation are involved.

SUMMARY:
This study assesses brain connectivity and function of individuals ages 13-25 at a prodromal or early stage of a psychotic disorder. Participation involves approximately 3 hours of MRI scanning and up to 6 hours of behavioral testing at Washington University School of Medicine's campus.

DETAILED DESCRIPTION:
Schizophrenia is a devastating illness inflicting about 1% of the population worldwide. Symptoms of schizophrenia include paranoia, hallucinations, and disorganized behaviors, and is associated with lifelong occupational and social disability. It typically develops in adolescence or early adulthood, which are particularly formative periods in life when major educational, vocational, and social life changes occur, and then the brain undergoes a rearrangement of critical neural circuits. The "prodrome" is the period before the onset of a psychotic disorder, like schizophrenia. Prodromal youth often have significant emotional distress and social withdrawal, and family members may observe a concerning change in behavior or school or work performance. Identifying those at clinical high risk for a psychotic disorder is important, as early intervention can improve symptoms and functioning, and could prevent the eventual development of a psychotic disorder. This study will focus on individuals aged 13-25 years who have met criteria for a psychosis-risk syndrome (or attenuated psychosis syndrome) or are at a very early stage (first 3 years after diagnosis) of a psychotic disorder, such as schizophrenia or schizoaffective disorder. Involvement will be either 2 or 3 partial days at Washington University and will involve approximately 3 hours of MRI scanning and up to 6 hours of behavioral testing. Additionally, the investigators will study the effect of genetics on the patterns of brain connectivity in various psychiatric populations. DNA will be collected non-invasively from saliva and stored and processed in Washington University facilities.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 13 and 25
* Meet diagnostic criteria for a prodromal syndrome or early psychosis by either meeting: 1) criteria for psychosis-risk on the structured assessment of psychosis-risk syndrome, or 2) meeting criteria for a psychotic disorder on the SCID diagnostic interview only within the last 3 years.
* Understand and sign an informed consent (or assent form for minors) document in English

Exclusion Criteria:

* IQ of 70 or under
* Past or current history of clinically significant central nervous system disorder that may contribute to psychotic symptoms or confound their assessment
* Pregnancy
* The diagnostic symptoms are clearly caused by an Axis I disorder, including substance use disorders, as judged by the evaluating clinician.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals aged 13-25 years who have met criteria for a psychosis-risk syndrome or at a very early stage of a psychotic disorder, such as schizophrenia or schizoaffective disorder.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-19 (Estimated); Study Completion 2021-06-19 (Estimated)

PRIMARY OUTCOMES:
MRI Brain Imaging | within one month of study enrollment
  The current project aims to uncover latent, homogenous, connectivity phenotypes using neuroimaging tools, which are free from the limitations of traditional diagnostic boundaries, and which correlate with clinical characteristics. The investigator will use resting state functional connectivity MRI (rs-fcMRI), diffusion MRI (dMRI) and tract-based spatial statistics (TBSS) to identify brain signatures that cut across psychotic disorders, including schizophrenia.

SECONDARY OUTCOMES:
DNA testing through saliva | within one month of study enrollment
  Saliva samples will be collected from participants for DNA extraction and the development of lymphoblastoid cell lines. DNA is used for research purposes only, for studies assessing brain connectivity.

OTHER OUTCOMES:
Hair sample for cortisol measurement | within one month of study enrollment
  To see how cortisol levels can help characterize brain imaging findings

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States